CLINICAL TRIAL: NCT04138875
Title: A Phase II Multicenter Open Label Risk Stratified Sequential Treatment With Rituximab, Brentuximab Vedotin and Bendamustine (RBvB) in Patients Newly Diagnosed.
Brief Title: A Risk Stratified Sequential Treatment With Rituximab, Brentuximab Vedotin and Bendamustine (RBvB)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, FRANCESCA MONTANARI, Assistant Professor of Medicine, Yale University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2000029609
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: PTLD; Lymphoid Tumor; Hematopoietic/Lymphoid Cancer; Plasmacytic Hyperplasia PTLD; Infectious Mononucleosis; Florid Follicular Hyperplasia PTLD; Polymorphic PTLD; Monomorphic PTLD; Classical Hodgkin Lymphoma Type PTLD
MeSH Terms: conditions — Hematologic Neoplasms; Infectious Mononucleosis | interventions — Rituximab; Brentuximab Vedotin; Bendamustine Hydrochloride

STUDY DESIGN:
Intervention Model Description: This is an open label, sequential, risk stratified study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low Risk (Active Comparator): Low risk patients (those in complete response (CR) after induction) will receive rituximab (375mg/m2) and brentuximab vedotin (1.8mg/m2) on day 1 of 21 day cycles, for 4 cycles.
  Interventions: Drug: Rituximab; Drug: Brentuximab Vedotin
- High Risk (Active Comparator): High risk patients (those who do not achieve a CR after induction), will receive rituximab (375mg/m2) and brentuximab vedotin (1.8mg/m2) on day 1 and bendamustine (90mg/m2) on day 1-2 of 21 day cycles for up to 8 cycles. Interim imaging will be performed in cycle 4 (days 14-21) and patients achieving CR will receive additional 2 cycles for a total of 6, patients achieving partial response (PR) will receive 4 additional cycles.
  Interventions: Drug: Rituximab; Drug: Brentuximab Vedotin; Drug: Bendamustine

INTERVENTIONS:
Drug: Rituximab — Rituximab is dosed at 375mg/m2 as an intravenous infusion. No adjustments are necessary for hepatic or renal impairment. Dosing will be done on baseline weight and height, however in patients who experience a >10% change in weight dosing will be readjusted.
  Other Names: Rituxan
Drug: Brentuximab Vedotin — Brentuximab vedotin is to be given as intravenous infusion at a dose of 1.2mg/kg during induction and 1.8mg/kg with each cycle. Dose reductions to 1.2mg/kg are allowed at investigator discretion.
  Other Names: Adcetris
Drug: Bendamustine — Bendamustine is to be given intravenously at a dose of 90mg/m2 on day 1 and day 2 of each high risk cycle. Dose reductions to 60mg/m2 are allowed at investigator discretion.
  Other Names: Bendamustine hydrochloride
  Arms: High Risk

SUMMARY:
This is an open label, risk-stratified, sequential treatment, phase 2 study of newly diagnosed post-transplant lymphoproliferative disorders with positive CD20 and CD30 expression. It includes an induction phase with rituximab and brentuximab vedotin (RBv), followed by a treatment phase with RBv or RBv in combination with bendamustine (RBvB) based on response to induction.

The primary end point is treatment efficacy measured as the overall response rate (ORR) and progression free survival (PFS).

DETAILED DESCRIPTION:
Post-Transplant Lymphoproliferative Disorders (PTLD) are defined by the revised 2017 edition of the WHO Classification of Tumours of Haematopoietic and Lymphoid Tissues as "lymphoid or plasmacytic proliferations that develop as a consequence of immunosuppression in a recipient of a solid organ, bone marrow or stem cell allograft". Within this definition 4 distinct categories exist, including: (1) Non-destructive PTLDs (plasmacytic hyperplasia, infectious mononucleosis, and florid follicular hyperplasia) (2) Polymorphic PTLD; (3) Monomorphic PTLD and (4) Classical Hodgkin Lymphoma type PTLD.

The incidence of PTLD varies between different transplanted organs. Across all transplants monomorphic PTLD is the most common accounting for 75% of all cases. Lymphoma derived of B- cell origin account for the majority of cases (70%), while T-cell neoplasms represent a small minority (5%). Within monomorphic PTLD 50% of cases demonstrate association with the Epstein Barr Virus (EBV). Polymorphic PTLD accounts for 15-20% of all PTLD cases with the majority demonstrating EBV involvement. Early lesions account for 5% of PTLD and are all uniformly associated with EBV as are all the cases of Classic Hodgkin Lymphoma type PTLD.

The current understanding of the pathogenesis of PTLD is incomplete. Despite concerted efforts, the investigators are unable to predict who will develop PTLD and do not understand why only 1 - 2% of all transplant recipients develop these disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 70 at the time of signing informed consent
2. Patient must have histologically confirmed newly diagnosed polymorphic or monomorphic PTLD defined according to the 2016 World Health Organization (WHO) classification criteria.
3. Diagnostic archival tissue available for review and correlative studies
4. Previous solid organ or allogeneic hematopoietic stem cell transplant
5. Measurable disease
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
7. Patients must have adequate organ and marrow function
8. Negative urine or serum pregnancy test for women of childbearing potential
9. Patients must be able to understand and to sign a written consent document.

Exclusion Criteria:

1. Previous treatment for PTLD with the exception of immunosuppression reduction
2. Known involvement of the central nervous system by the PTLD
3. Known allergic reactions against foreign proteins
4. Uncontrolled inter-current illness including active infection, acute graft versus host disease and/or transplant organ rejection
5. Active concurrent malignancy with the exception of non-melanoma skin cancer, carcinoma in situ of the cervix or localized prostate cancer
6. Severe non-compensated diabetes mellitus
7. Pre-existing neuropathy grade 2 or greater
8. Pregnant or lactating
9. Psychiatric illness / social situations that would limit compliance with study requirements
10. Patients with previous hypersensitivity to Rituximab
11. Known HIV positive.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) (complete + partial response rate) | Up to 84 days of treatment (4 cycles of treatment)
  Overall response rate (ORR) (complete + partial response rate) of the combination of rituximab, brentuximab vedotin +/-bendamustine in patients.
Progression free survival (PFS) rate | Up to 84 days of treatment (4 cycles of treatment)
  Progression free survival (PFS) of the combination of rituximab, brentuximab vedotin +/-bendamustine in patients.

SECONDARY OUTCOMES:
ORR at the end of the induction phase | Up to 126 days of treatment (6 cycles of treatment)
  ORR at the end of the induction phase with rituximab and brentuximab vedotin (RBv) in patients
Duration of response (DOR) | Up to 84 days of treatment (4 cycles of treatment)
  duration of response (DOR) of the combination of rituximab, brentuximab vedotin +/-bendamustine in patients with newly diagnosed polymorphic and monomorphic CD20+ and CD 30+ PTLD.
Overall survival (OS) | 3 years
  Overall survival (OS) of the combination of rituximab, brentuximab vedotin +/-bendamustine in patients with newly diagnosed polymorphic and monomorphic CD20+ and CD 30+ PTLD

CONTACTS AND LOCATIONS:
Overall Officials: Francesa Montanari, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No